CLINICAL TRIAL: NCT02658448
Title: GTx-024 as a Treatment for Stress Urinary Incontinence in Women: A Proof of Concept Study
Brief Title: GTx-024 as a Treatment for Stress Urinary Incontinence in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G201001
Record Dates: First submitted 2016-01-13; First posted 2016-01-18 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — ostarine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GTx-024 3 mg (Experimental): GTx-024 softgel capsules will be administered once daily to a total dose of 3 mg for up to 12 weeks.
  Interventions: Drug: GTx-024

INTERVENTIONS:
Drug: GTx-024 — GTx-024 softgel capsules will be administered once-daily to a total dose of 3 mg
  Other Names: enobosarm

SUMMARY:
The purpose of this study is to determine whether GTx-024 is safe and effective in the treatment of stress urinary incontinence in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary, written and signed, informed consent
* Female
* Age18 to 80 years old be clinically confirmed as postmenopausal. Subjects must have undergone the onset of spontaneous, medically induced or surgical menopause prior to the start of this study. Spontaneous menopause is defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
* SUI symptoms for at least 6 months duration
* Predominant SUI (MESA questionnaire)
* 24 hour pad weight >3 gms at baseline
* A minimum of 1 SUI episode per day, in the 3 day diary
* 3-15 SUI episodes per day, averaged over 3 days, in the 3 day diary
* Serum AST and ALT within normal limits
* Total bilirubin within normal limits
* Positive Bladder Stress Test during screening
* Subject agrees to not start any new treatment (medication or otherwise) that is known to affect lower urinary tract function throughout the treatment and follow up periods
* Subject agrees to maintain on a stable dose of any medication known to affect lower urinary tract function, including but not limited to anticholinergics, tricyclic antidepressants, or alpha-adrenergic blockers, throughout the treatment and follow-up period

Exclusion Criteria:

* Pelvic floor physical therapy in a clinical setting within 30 days prior to screening
* History of pelvic radiation treatment
* History of urethral diverticula
* History of urethral sling, anterior prolapse repair, ureteral bulking agents and/or other SUI procedure or surgery
* Known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant urological findings, including pelvic floor abnormalities which, in the judgement of the investigator, could impact treatment
* Urinary incontinence of neurogenic etilogy
* Patient is morbidly obese (defined as 100 pounds over their ideal body weight, or body mass index 40 or greater)
* Chronic hepatitis
* Hepatic cirrhosis
* HIV and/or hepatitis A, B, or C
* Subjects taking systemic hormone products
* Subjects with a history of breast or endometrial cancer
* Myocardial infarction or arterial thromboembolic events within 6 months prior to Baseline, severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, serious uncontrolled cardiac arrhythmia grade II or higher according to NYHA, uncontrolled hypertension (systolic > 150 and/or diastolic > 100 mm Hg)
* Subjects with an entry measurement of > 5 mm endometrial stripe thickness
* Clinically confirmed urinary tract infection
* Any other condition which per investigators' judgment may increase subject risk

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M. Peters, MD, Principal Investigator — Corewell Health East
Locations (3):
- United States (3):
  - William Beaumont Hospital, Royal Oak, Michigan
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Penn Center for Continence and Pelvic Health, University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GTx-024 3 mg
Started | 19
Completed | 18 (One patient was lost to follow-up after enrollment and prior to visit 1)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | GTx-024 3 mg
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 61.4 [45 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Baseline mean number of stress leaks per day [Mean (Full Range); unit: number of leaks per day] | 5.17 [3.33 to 10.33]

OUTCOME MEASURES:

1. Primary Outcome: The Mean Percent Change in Number of Stress Incontinence Episodes/Day as Assessed by Patient Completion of the 3 Day Voiding Diary
Description: To describe the effect of 12 weeks of treatment of GTx-024 on the number of stress incontinence episodes/day as assessed by patient completion of the 3 day voiding diary
Time Frame: 12 weeks
Population: all patients with at least one post enrollment assessment
Measure: Mean (Full Range); unit: percent reduction
Arm/Group | GTx-024 3 mg
Number analyzed (Participants) | 18
percent reduction | 81 [50 to 100]

2. Secondary Outcome: Stress Urinary Incontinence as Assessed by 24 Hour Pad Weight Test. Mean Percent Change in Pad Weight
Description: To describe the effect of 12 weeks of treatment of GTx-024 on SUI as assessed by 24 hour pad weight test. Mean percent reduction in pad weight
Time Frame: 12 weeks
Population: all patients with at least one post enrollment assessment
Measure: Mean (Full Range); unit: percent
Arm/Group | GTx-024 3 mg
Number analyzed (Participants) | 18
percent | 71 [27 to 126]

3. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: To describe the safety profile of GTx-024 3 mg PO daily in subjects with stress urinary incontinence.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GTx-024 3 mg
Number analyzed (Participants) | 19
Participants | 9

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | GTx-024 3 mg
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTx-024 3 mg (N=19)
headache (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
hot flash (Endocrine disorders) | 1 (1)
insomnia (General disorders) | 1 (1)
urinary frequency (Renal and urinary disorders) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
tooth abscess (Infections and infestations) | 1 (1)
vaginal itching (Reproductive system and breast disorders) | 1 (1)
vaginal bleeding (Reproductive system and breast disorders) | 1 (1)
elevated alanine aminotransferase (Investigations) | 1 (1)
low HDL (Investigations) | 1 (1)
elevated HDL (Investigations) | 1 (1)
low sex hormone binding globulin (Investigations) | 1 (1)
breast cyst (Reproductive system and breast disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
proteinuria (Renal and urinary disorders) | 1 (1)
ketonuria (Renal and urinary disorders) | 1 (1)
bilirubinuria (Renal and urinary disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
pelvic floor muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1)
periodontitis (Infections and infestations) | 1 (1)
thrush (Infections and infestations) | 1 (1)
cold (Infections and infestations) | 1 (1)
flu (Infections and infestations) | 1 (1)
abdominal muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (1)
elevated INR (Investigations) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
cyctocele (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open label, small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT02658448/Prot_SAP_000.pdf